CLINICAL TRIAL: NCT03994692
Title: Evaluation of Patient Satisfaction Using Autogenous Inlay (Sandwich) Eminoplasty Versus Patient Specific Poly Ether-ether Ketone (PEEK) Onlay Implant in Treatment of Chronic Condylar Dislocation A Randomized Control Trial
Brief Title: Evaluation of Patient Satisfaction Using Autogenous Inlay (Sandwich) Eminoplasty Versus Patient Specific Poly Ether-ether Ketone (PEEK) Onlay Implant
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Collaborators: El-Galaa Military Medical Complex (Other Government)
Responsible Party: Principal Investigator, mustafa gamal abdel kawy, resident of oral & maxillofacial surgery department, El-Galaa Military Medical Complex
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: omfs 3-3-3
Record Dates: First submitted 2019-06-19; First posted 2019-06-21 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Mandibular Dislocation
Keywords: PEEK eminoplasty ,autogenous inlay (sandwich) eminoplasty

STUDY DESIGN:
Intervention Model Description: * randomized control trial
  * trials will be carried out in hospital of oral & maxillofacial department at faculty of oral and dental medicine of Cairo university
  * equal randomization participants with equal probabilities for intervention
  * positive controlled , both groups receiving treatment
  * parallel group study , each group of patient receive single treatment simultaneously
Masking Description: because the two intervention in this trial are clearly different and easily recognized by participant and investigator , neither investigators nor participant can be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEEK eminoplasty (Experimental): CT scan with bony window for facial bones and DICOM files on CD .then, Using cad cam software (mimics 15) , the virtual design and surgery will be done.
  under general anathesia The TMJ will be exposed using the endural incision line and the articular eminence will be identified then blunt dissection so that the front wall of the articular capsule can be exposed completely.
  * The patient specific PEEK eminence will be inserted and secured with two to three pre-planed screws .
  * Functional mandibular movements were reproduced to confirm absence of subluxation and then closure
  Interventions: Device: PEEK eminoplasty
- autogenous onlay grafting eminoplasty (Active Comparator): under general anesthesia , chin graft was taken Layered Endural approach to TMJ making wedge in eminence by mallet & chisel (green stick fracture), then wedging piece of chin graft to increase the height of the eminence creating an obstacle to treat dislocation by manipulation of patient mandible intra operative.
  - Functional mandibular movements were reproduced to confirm absence of subluxation then closure
  Interventions: Procedure: autogenous onlay grafting eminoplasty

INTERVENTIONS:
Device: PEEK eminoplasty — making obstacle at eminence using patient specefic PEEK device
  Other Names: poly ether - ether ketone
  Arms: PEEK eminoplasty
Procedure: autogenous onlay grafting eminoplasty — making obstacle at eminence using chin graft
  Other Names: grafting eminoplasty
  Arms: autogenous onlay grafting eminoplasty

SUMMARY:
Aim of the study:

The aim is minimize morbidity in treatment of TMJ dislocation. Hypothesis: Alternate hypothesis that treatment tmj dislocation with PEEK eminoplasty will be more efficient than using autogenous inlay technique

PICO:

Problem (P): patients with un pleasant painful dislocated tmj Intervention (I): eminoplasty with patient specific poly ether-ether ketone (PEEK) onlay implant Control Group (C): autogenous inlay (sandwich) eminoplasty Outcome (O): patient Satisfaction, dislocation treatment (normal range of mouth opening), less morbidity.

DETAILED DESCRIPTION:
Aim of the study:

The aim is minimize morbidity in treatment of TMJ dislocation. Hypothesis: Alternate hypothesis that treatment tmj dislocation with PEEK eminoplasty will be more efficient than using autogenous inlay technique

PICO:

Problem (P): patients with un pleasant painful dislocated tmj Intervention (I): eminoplasty with patient specific poly ether-ether ketone (PEEK) onlay implant Control Group (C): autogenous inlay (sandwich) eminoplasty Outcome (O): patient Satisfaction, dislocation treatment (normal range of mouth opening), less morbidity.

8. Trial design: Type: Parallel, two arm, randomized clinical trial. Allocation ratio: 1:1 Superiority framework

III. Methods A) Participants, interventions & outcomes 9. Study settings: Diagnosis in outpatient clinic of Oral and Maxillofacial surgery at the faculty of dentistry, Cairo University, Urban area, Cairo Governorate, Egypt.

The surgery will be in O.R rooms or in the outpatient clinic of the same faculty.

11. Interventions

Control Group:

Patient preparation The operation can be performed under general anesthesia. mental nerve blocks will be given and infiltration for hemostasis.

After allowing adequate time for vasoconstrictor effects to take place, the incision is initiated in a layered approach through the labial mucosa and is continued through the mentalis muscles and periosteum.

Exposure of the symphyseal bone is undertaken using periosteal elevators and the mental nerves are visualized bilaterally.

The roots of the incisors and canines should be localized and bone cuts should be made at least 5 mm inferior to the root apices.

The roots of canines can impede the operation and limit the size of graft. Similarly, the surgeon should stay at least 5 mm away from the inferior border of the symphysis and the mental foramina.

Bone cuts can be made with a bur or reciprocating saw under copious saline irrigation. When the desired bone cuts have been completed, thin straight or curved osteotomes are then used to deliver the graft Hemostasis can be achieved using resorbable hemostatic agents or fibrin glue. Long-lasting local anesthetic, e.g. bupivacaine, can be applied to the area to achieve longer analgesia.

The wound closure is done in two layers with a resorbable suture for the muscle layer and fast-resorbing suture for the mucosa.

Flexible skin tape can be used on the chin for 3-5 days to reduce swelling and prevent wound dehiscence.

Layered Endural approach to TMJ making wedge in eminence by mallet & chisel (green stick fracture), then wedging piece of chin graft to increase the height of the eminence creating an obstacle to treat dislocation by manipulation of patient mandible intra operative.

* Functional mandibular movements were reproduced to confirm absence of subluxation and checked for interference and any required adjustments made.
* A multilayer closure of the incisions will be accomplished using Vicryl sutures (88).

Intervention group ; CT scan will be done with the following criteria;

bony window for facial bones, axial cuts, minimal slice thickness, minimal intervals between the cuts, guantry tilt equals zero and finally DICOM files on CD .then, Using cad cam software (mimics 15) , the virtual design and surgery will be done.

Patient Preparation;

* All surgeries will be performed under general anaesthesia (naso-endotracheal intubation)
* Then the entire periarticular region and overlying skin will be infiltrated by 2% lidocaine (20 ml lidocaine + adrenalin 1%) via a 25 gauge needle as an additional anaesthesia.
* Benzyl penicillin 2 MIU in combination with dicloxacillin 1 g will be administered intravenously as prophylactic antibiotics.
* A line is drawn between the lateral eyebrow and tragus. The articular fossa and condylar head is located 10 mm anterior to the tragus and 2-5 mm below this line.
* The temporofacial branch has relatively a constant course and vector being on a line located 0.5 cm below the tragus of the ear, in the direction of the eyebrow and passing 1.5 cm above the lateral eyebrow. Just anterior to the condylar head where the articular eminence will be identified by palpation and marked.

The TMJ will be exposed using the endural incision line and the articular eminence will be identified

* To locate the articular eminence precisely, tissue must be exposed layer by layer until the articular eminence is located. Then, a tunnel will be formed using blunt dissection so that the front wall of the articular capsule can be exposed completely.(89-90-91 )
* The patient specific PEEK eminence will be inserted and secured with two to three pre-planed screws .
* Functional mandibular movements were reproduced to confirm absence of subluxation and checked for interference and any required adjustments made.
* A multilayer closure of the incisions will be accomplished using Vicryl sutures.

For both groups masseter muscle scarification through intra oral approach will be done with post-operative intermaxillary fixation using ivy loops

Post-operative instructions:

According to Oral Maxillo-fac Surg Clin North Am (Quinn PD, 2000):

The following postoperative protocol will be used for patients of both groups:

* Broad-spectrum antibiotics (penicillin V 1 g, or clindamycin 600 mg) and non-steroidal anti-inflammatory drugs (NSAIDS) will be prescribed for 1 week.
* The patients will be told to stay on a soft diet for 5 days and encouraged to resume a normal diet as soon as possible.
* Physiotherapy will start on postoperative day 1, and patients will be encouraged to increase the exercise program as soon as possible.
* Patients will be advised to continue physiotherapy for at least 1 year and possibly longer.
* Cone Beam CT (CBCT) imaging will be performed at the first follow-up visit in order to visualize the position of the patient specific titanium eminence, as well as the position of the retention screws and their relationships to the surrounding vital structures following surgery.

Visit: (every month till 4 month after operation) For group I: Regular follow up with measuring maximum inter incisal distance with a caliper , check normal mandibular movement & other problems like pain ,discomfort & swelling For group II: Regular follow up with measuring maximum inter incisal distance with a caliper , check normal mandibular movement & other problems like pain ,discomfort & swelling

ELIGIBILITY:
Inclusion Criteria:

* - Patient with recurrent dislocation with maximum inter incisal opening over 55mm
* Long-standing dislocation of the TMJ involving both fixation for more than 3 weeks and the failure of manual reduction
* Failure of conservative strategies such as orientation to self-limit jaw movement and the use of a chin-cap or bandage
* Both sexes
* Age between 18 and 48 years.
* Highly motivated patients.

Exclusion Criteria:

* Post-menopausal females with osteoporosis
* Patient with uncontrolled systemic disease
* pregnancy
* psychological disorders, drug or alcohol dependency
* Known allergies or sensitivities to dental materials, including PEEK, Titanium or general anesthetic agents
* Inability to return for follow up visits.
* Refusal of participation from the patient

Ages: 22 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Estimated)
Dates: Start 2019-06-20 (Estimated); Primary Completion 2020-07-20 (Estimated); Study Completion 2021-03-20 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction: Question | up to 4 month after operation
  Questioning the patient about if there is any dislocation or any limitation to mandibular movement

SECONDARY OUTCOMES:
Maximal Incisal Opening | follow up for 4 month
  measured with Caliper
Intra operative time | during operation
  measured with time calculation
Post operative pain: VAS | follow up for 2 weeks up to 4 month
  measured with visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: mohamed mounir, Phd, Study Director — faculty of oral and dental medecine cairo university

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1-Mayer L. Recurrent dislocation of the jaw. J Bone Joint Surg1933;15:22Y25 2- Van der Kwast WA. Surgical management of bilateral habitual luxation of the mandible. Int J Oral Surg 1978;7:329Y332 3- Gosserez M, Dautrey J. Osteoplastic bearing for the treatment of temporomandibular luxations. In: Oral Surgery Transactions of 2nd Congress of Int Assoc Oral Surg Copenhagen. 1967:261Y264 4- Lindemann A. Die chirurgische behandlung der erkrankungen des kiefergelenkes. Z Stoma 1925;23:395Y 406 5- Iizuka T, HNdaka H, Murakami K, et al. Chronic recurrent anterior luxation of the mandible. Int J Oral Maxillofac Surg 1988; 17:170Y172